CLINICAL TRIAL: NCT00694083
Title: A Phase I Study of MK-8669 in Patients With Metastatic or Locally Advanced Solid Tumors
Brief Title: Study of Ridaforolimus (MK-8669) in Participants With Solid Tumors (MK-8669-003)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8669-003; 2008_011 (Other: Study Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-10 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — ridaforolimus

ARMS (1):
- Ridaforolimus (Experimental): Ridaforolimus (MK-8669), 20 or 40 mg administered orally on Day 1 followed by a washout of at least 6 days, then QD x5 (five consecutive days) followed by a 2-day holiday through Day 28 (Cycle 1), and QD x5 followed by a 2-day holiday for 21 days (Cycle 2 and subsequent cycles).
  Interventions: Drug: Ridaforolimus

INTERVENTIONS:
Drug: Ridaforolimus — Ridaforolimus (MK-8669), 20 or 40 mg administered orally on Day 1 followed by a washout of at least 6 days, then QD x5 (five consecutive days) followed by a 2-day holiday through Day 28 (Cycle 1), and QD x5 followed by a 2-day holiday for 21 days (Cycle 2 and subsequent cycles)
  Other Names: MK-8669

SUMMARY:
A clinical study evaluates the safety, tolerability, and pharmacokinetics of ridaforolimus (MK-8669) in participants with locally advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically - Or Cytologically- Confirmed Metastatic Or Locally Advanced Solid Tumors That Have Failed To Respond To Standard Therapy, Or For Which Adequate Standard Therapy Does Not Exist
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Adequate Organ Function

Exclusion Criteria:

* Participant Who Has Had Chemotherapy, Radiotherapy, Or Biological Therapy Within 4 Weeks (6 Weeks For Nitrosoureas Or Mitomycin C) Prior To Registration
* Any central nervous system Metastasis Which Has Symptoms Or Requires Treatment
* Any Primary Central Nervous System Tumor
* Any Symptomatic Ascites Or Plural Effusion Which Requires Treatment
* A History Or Current Evidence Of Any Clinically Significant Disease That Might Confound The Results Of The Study, Complicate The Interpretation Of The Study Results, Interfere With The Participant's Participation, Or Pose An Additional Risk To The Participant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06-10 (Actual); Primary Completion 2009-09-06 (Actual); Study Completion 2009-09-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Ridaforolimus Dose Limiting Toxicities | Cycle 1 (28 days)

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve (AUC) for Ridaforolimus for Day 1 (Single Dose, 20 mg or 40 mg) | Day 1
Area Under the Plasma Concentration-Time Curve (AUC) for Ridaforolimus for Day 26 (Multiple Doses, 20 mg or 40 mg) | Day 26
Maximum Plasma Concentration (Cmax) for Day 1 (Single Dose of Ridaforolimus, 20 mg or 40 mg) | Day 1
Maximum Plasma Concentration (Cmax) for Day 26 (Multiple Doses of Ridaforolimus, 20 mg and 40 mg) | Day 26

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Seki Y, Yamamoto N, Tamura Y, Goto Y, Shibata T, Tanioka M, Asahina H, Nokihara H, Yamada Y, Shimamoto T, Noguchi K, Tamura T. Phase I study for ridaforolimus, an oral mTOR inhibitor, in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2012 Apr;69(4):1099-105. doi: 10.1007/s00280-011-1788-4. Epub 2011 Dec 6. PMID 22143378